CLINICAL TRIAL: NCT01976000
Title: The Impact of Preoperative Knowledge of the Colonic Vascular Anatomy on the Learning Curve for Laparoscopic Colorectal Resection
Brief Title: Influence of CT 3D on the Learning Curve of Laparoscopic Colorectal Resection
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Saverio Mari, MD, University of Roma La Sapienza
Other Study IDs: DS-009
Record Dates: First submitted 2013-10-29; First posted 2013-11-05 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2014-02

CONDITIONS: Learning Curve of Laparoscopic Colorectal Resections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: the surgeons were able to view 3D reconstructions before and during surgery
  Interventions: Procedure: multi-slice Computed Tomography angiography and three-dimensional reconstruction software
- Group B: the surgeons were only able to view 3D reconstructions after the surgery

INTERVENTIONS:
Procedure: multi-slice Computed Tomography angiography and three-dimensional reconstruction software
  Groups: Group A

SUMMARY:
Laparoscopic colorectal surgery has been widely accepted worldwide; however, despite the well-known benefits and comparable oncological outcomes, it is still limited by a lack of tactile sensation and a reduced operative field view. In addition, the inconsistency in the number and course of the mesenteric vessels significantly influences the learning curve with 30 to 70 cases required for proficiency. To overcome these limitations, the vascular anatomy can be mapped using CT-angiography, and the images can be processed with rendering software to reconstruct a three-dimensional model of the mesenteric vessels. The aim of this study was to assess the influence of visualizing the three-dimensional vascular anatomy on the learning curve for laparoscopic colorectal surgery.All patients who underwent laparoscopic left or right hemicolectomies between January 2012 and January 2014 were evaluated for inclusion in this study. To assess the influence of preliminary knowledge of colonic vascular anatomy on the learning curve, we considered 2 groups of two surgeons with different levels of experience. In the first group (group A), the surgeons were able to view 3D reconstructions before and during the surgery, while the surgeons in Group B were only able to view the 3D reconstructions after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients in which standard laparoscopic right or left hemicolectomy was planned

Exclusion Criteria:

* patients who underwent extended right hemicolectomy and segmental colectomy or sigmoidectomy and patients for whom the surgical technique was modified intraoperatively
* patients who underwent anterior rectal resection and emergency procedures for complicated diverticulitis were excluded because these procedures require higher technical skills.
* Patients who had an ASA score of IV, a BMI over 40 or contraindications for laparoscopy were also excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We included only patients in which standard laparoscopic right or left hemicolectomy was planned and who needed a CT scan but had not received a scan prior to their first office visit.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
operating time | operating time

SECONDARY OUTCOMES:
intraoperative and postoperative complications | first 2 week after surgery
hospital stay | first 2 weeks after surgery
oncological clearance | first 2 weeks after surgery
  radicality and number of harvested lymph nodes

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Sant'Andrea, Rome, Italy